CLINICAL TRIAL: NCT03620890
Title: Detemir Versus NPH for Type 2 Diabetes Mellitus in Pregnancy: a Comparative-effectiveness, Open Label, Randomized Controlled Trial
Brief Title: Detemir Versus NPH for Type 2 Diabetes Mellitus in Pregnancy
Acronym: Determin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Michal Fishel Bartal, Assistant Professor of OB GYN, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0575
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin, Isophane; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neutral Protamine Hagedorn (NPH) (Active Comparator): NPH will peak between 4-12 hours after injection with a duration of action around 14 hours
  Interventions: Drug: Neutral Protamine Hagedorn (NPH)
- Detemir (Active Comparator): Detemir is characterized by a gentle rise and fall with a longer duration of action (18-20 hours)
  Interventions: Drug: Detemir insulin

INTERVENTIONS:
Drug: Neutral Protamine Hagedorn (NPH) — NPH will peak between 4-12 hours after injection with a duration of action around 14 hours
  Arms: Neutral Protamine Hagedorn (NPH)
Drug: Detemir insulin — Detemir is characterized by a gentle rise and fall with a longer duration of action (18-20 hours)
  Arms: Detemir

SUMMARY:
To determine whether use of detemir compared to neutral protamine hagedorn (NPH) decreases rates of composite neonatal outcome and maternal hypoglycemia events in women with Type 2 Diabetes Mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Preexisting type 2 diabetes mellitus requiring medical treatment or
* overt diabetes diagnosed prior to 20 weeks of gestation using either Hemoglobin A1c (HBA1C) ≥ 6.5 or fasting glucose ≥126 mg/dl or random blood glucose ≥ 200 mg/dl or two step method ( 50g glucose challenge test (GCT) >135 mg/dl followed by 100 GCT with at least 2 values above thresholds: Fasting Blood Glucose (FBG) >90, 1 hr >180, 2 hr > 155, 3 hr > 140 mg/dl).
* Gestational age ≤20 weeks
* Willing to start insulin therapy or to continue insulin treatment during pregnancy
* Singleton or twin pregnancy

Exclusion Criteria:

* Known allergy/prior adverse reaction to NPH/detemir
* Patients <18y
* Known major fetal anomalies
* Diabetic nephropathy (Creatinine (Cr)≥1.5)
* Diabetic proliferative retinopathy
* Patients with Type 1 diabetes or gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fishel Bartal, MD, Principal Investigator — University of Texas Health Science Center of Houston
Locations (1):
- University of Texas Health Science Center of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fishel Bartal M, Ward C, Blackwell SC, Ashby Cornthwaite JA, Zhang C, Refuerzo JS, Pedroza C, Lee KH, Chauhan SP, Sibai BM. Detemir vs neutral protamine Hagedorn insulin for diabetes mellitus in pregnancy: a comparative effectiveness, randomized controlled trial. Am J Obstet Gynecol. 2021 Jul;225(1):87.e1-87.e10. doi: 10.1016/j.ajog.2021.04.223. Epub 2021 Apr 15. PMID 33865836

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Started | 57 | 51
First Trimester Miscarriage | 2 | 1
Major Fetal Anomalies (Hypoplastic Left Heart and Sacral Agenesis) With 2nd Trimester Stillbirth | 1 | 0
Major Fetal Anomaly (Holoprosencephaly) With 2nd Trimester Pregnancy Termination | 1 | 0
Completed | 53 | 50
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH) | Total
Number analyzed (Participants) | 57 | 51 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 51 | 108
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (6.2) | 32.5 (6.0) | 32.3 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 51 | 108
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 0 | 4
  Hispanic | 36 | 31 | 67
  Non-Hispanic Black | 14 | 14 | 28
  Non-Hispanic White | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 51 | 108
Number of maternal participants who had private insurance for prenatal care [Count of Participants; unit: Participants] | 22 | 18 | 40
Number of maternal participants who were nulliparous [Count of Participants; unit: Participants] — Nulliparous means never given birth before.
  Participants | 5 | 7 | 12
Number of maternal participants with body mass index (BMI) greater than 30 [Count of Participants; unit: Participants] | 51 | 38 | 89
Number of maternal participants with diabetes mellitus diagnosed before pregnancy [Count of Participants; unit: Participants] | 44 | 42 | 86
Number of maternal participants with HbA1c level greater than 6.5% [Count of Participants; unit: Participants] — HbA1c level is percentage of red blood cells (RBCs) that have sugar attached to hemoglobin (Hb).
  Participants | 37 | 34 | 71
Number of maternal participants with chronic hypertension [Count of Participants; unit: Participants] | 12 | 17 | 29
Number of maternal participants with depression or anxiety [Count of Participants; unit: Participants] | 7 | 9 | 16
Number of maternal participants with thyroid disease [Count of Participants; unit: Participants] | 2 | 4 | 6
Number of maternal participants who smoked during pregnancy [Count of Participants; unit: Participants] | 2 | 0 | 2
Number of maternal participants who used alcohol during pregnancy [Count of Participants; unit: Participants] | 2 | 0 | 2
Number of maternal participants who used substances during pregnancy [Count of Participants; unit: Participants] | 3 | 1 | 4
Number of maternal participants who used rapid- or short-acting insulin [Count of Participants; unit: Participants] | 38 | 41 | 79
Number of maternal participants who used aspirin during pregnancy [Count of Participants; unit: Participants] | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Neonates With Composite Adverse Neonatal Outcome
Description: Composite Adverse Neonatal Outcome includes 1 or more of any of the following:
  * Neonatal intensive care unit (NICU) admission or
  * Neonatal hypoglycemia (<40 mg/dL in the first 24 hours of life and less than 50 mg/dL after) or requiring medical therapy or
  * Respiratory distress (need for at least 4 hours of respiratory support with supplemental oxygen, continuous positive airway pressure or ventilation at the first 24 hours of life or
  * Shoulder dystocia - defined as the need for any extra maneuvers, other than gentle downward traction of the fetal head in order to deliver the fetal body after the fetal head has been delivered or
  * Large for gestational age (LGA) -weight over 90th percentile of the expected value according to gestational age or
  * Macrosomia- Fetal weight above 4000g
Time Frame: From the time of delivery to the time of discharge (about 2-14 days)
Population: All participants had singleton pregnancies (that is, there were no twins).
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 31 | 35

2. Secondary Outcome: Maternal Mean Fasting Glucose
Time Frame: perinatal to postpartum (32 weeks)
Population: Data were not collected for this outcome measure.
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Maternal Mean Post Prandial Glucose
Time Frame: perinatal to postpartum (32 weeks)
Population: Data were not collected for this outcome measure.
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Maternal Subjects Who Experienced Hypoglycemic Events (<60 mg/dL) During Pregnancy
Time Frame: perinatal to postpartum (32 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 8 | 16

5. Secondary Outcome: Change in Maternal Weight During Pregnancy
Time Frame: perinatal to postpartum (32 weeks)
Measure: Median (Inter-Quartile Range); unit: kilograms (kg)
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
kilograms (kg) | 7.00 [1.00 to 12.00] | 9.00 [4.00 to 14.70]

6. Secondary Outcome: Number of Maternal Subjects Who Had Hypertensive Disorder During Pregnancy
Description: Hypertensive disorder includes gestational hypertension, preeclampsia, or superimposed preeclampsia.
Time Frame: perinatal to postpartum (32 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 22 | 27

7. Secondary Outcome: Number of Maternal Subjects Who Had Preeclampsia With Severe Features
Time Frame: perinatal to postpartum (32 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 12 | 16

8. Secondary Outcome: Number of Subjects Who Had Cesarean Delivery
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 32 | 30

9. Secondary Outcome: Number of Subjects Who Had Operative Vaginal Delivery
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 1 | 0

10. Secondary Outcome: Gestational Weeks at Delivery
Time Frame: at delivery
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
weeks | 37.10 [36.00 to 37.40] | 37.00 [34.10 to 37.40]

11. Secondary Outcome: Number of Neonates Who Where Small for Gestational Age (SGA)
Description: Small for gestational age (SGA) means that a fetus or an infant is smaller or less developed than normal for the baby's sex and gestational age. Small for gestational age (SGA) is defined as a birth weight that is below the 10th percentile.
Time Frame: at delivery
Population: All participants had singleton pregnancies (that is, there were no twins).
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 4 | 6

12. Secondary Outcome: Neonatal Hospital Admission Days
Time Frame: From the time of delivery to the time of discharge (about 2-14 days)
Population: All participants had singleton pregnancies (that is, there were no twins).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
days | 4.0 [2.0 to 8.0] | 4.1 [2.0 to 14.0]

13. Secondary Outcome: # of Neonates Who Had 5-minute Apgar Score < 7
Description: The Apgar score is determined by evaluating the newborn baby on each of five criteria (appearance, pulse, grimace, activity, respiration) on a scale from zero to two, then summing the five values obtained. The total score ranges from zero to 10. A higher score indicates a better outcome.
Time Frame: 5 minutes after delivery
Population: All participants had singleton pregnancies (that is, there were no twins).
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 3 | 2

14. Secondary Outcome: Number of Neonates Who Had Jaundice Requiring Therapy
Time Frame: From the time of delivery to the time of discharge (about 2-14 days)
Population: All participants had singleton pregnancies (that is, there were no twins).
Measure: Count of Participants; unit: Participants
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
Number analyzed (Participants) | 53 | 50
Participants | 15 | 11

ADVERSE EVENTS:
Time Frame: perinatal to postpartum (32 weeks)
Description: All deaths were pregnancy losses, and there were no maternal deaths.
Arm/Group | Detemir | Neutral Protamine Hagedorn (NPH)
All-Cause Mortality (participants affected / at risk) | 4/57 | 1/51
Serious Adverse Events (participants affected / at risk) | 16/57 | 10/51
Other Adverse Events (participants affected / at risk) | 0/53 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Detemir (N=57) | Neutral Protamine Hagedorn (NPH) (N=51)
First trimester miscarriage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Major fetal anomaly (holoprosencephaly) with termination of pregnancy in 2nd trimester (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Major fetal anomalies (hypoplastic left heart and sacral agenesis) with stillbirth in 2nd trimester (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Maternal admission to the hospital during pregnancy, other than admission for labor (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 8 (8)
Maternal readmission to hospital after delivery (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT03620890/Prot_SAP_000.pdf